CLINICAL TRIAL: NCT02884102
Title: Clinical-grade Molecular Profiling of Patients With Multiple Myeloma and Related Plasma Cell Malignancies
Brief Title: MMRF Molecular Profiling Protocol
Status: Active, not recruiting | Type: Observational
Sponsor: Multiple Myeloma Research Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MMRF-002
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2025-05-06 (Actual); Status verified 2023-02

CONDITIONS: Multiple Myeloma; Plasma Malignancy
Keywords: genetic sequencing; relapsed
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — bone marrow and peripheral blood samples will be obtained
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: genetic sequencing

SUMMARY:
This protocol is now being used as screening for the MyDRUG study

DETAILED DESCRIPTION:
Here we propose an "integrative sequencing approach" utilizing a 1500 gene exome comparative analysis between multiple myeloma or related plasma cell malignancies and normal cells coupled to capture transcriptome sequencing to provide a nearly comprehensive landscape of the genetic alterations for the purpose of identifying informative and/or actionable mutations in patients with multiple myeloma and plasma cell malignancies. The approach will enable the detection of point mutations, insertions/deletions, gene fusions and rearrangements, amplifications/deletions, and outlier expressed genes among other classes of alterations.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a diagnosis of multiple myeloma or related malignancy
2. Patients are undergoing standard of care bone marrow aspirates
3. Patients (male or female) from any race or ethnicity must be at least 18 years of age at the time of registration.
4. Procedure-specific signed informed consent form prior to initiation of any study-related procedures.

Exclusion Criteria:

1. It is the enrolling study physician's discretion to decide if a patient is not fit enough to undergo a bone marrow aspirate.
2. Patients who are incarcerated are not eligible to participate.
3. Women who are pregnant
4. Patients who have had another malignancy within the last five (5) years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix) where there is a possibility to contaminate the bone marrow aspirate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with multiple myeloma and other related disorders including, without limitation to, smoldering myeloma, monoclonal gammopathy of undetermined significance (MGUS), primary plasma cell leukemia, solitary plasmacytoma, and amyloidosis
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-06; Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
actionable mutations report | 10-14 days

SECONDARY OUTCOMES:
Survival Rates | Overall survival
Disease Recurrence | Time to Progression

CONTACTS AND LOCATIONS:
Overall Officials: Leif Bergsagel, M.D., Principal Investigator — Mayo Clinic
Locations (20):
- United States (19):
  - Mayo Clinic - Scottsdale, Scottsdale, Arizona
  - City of Hope, Duarte, California
  - UCSF Medical Center, San Francisco, California
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Ohio State University, Columbus, Ohio
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada